CLINICAL TRIAL: NCT06251219
Title: Active Case Finding of Clinical Hand Foot Mouth Disease in Children Aged 6 Months Old to 18 Years Old in Indonesia
Status: Not yet recruiting | Type: Observational
Sponsor: Sinovac Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: PRO-EV71/CA16-5002
Record Dates: First submitted 2024-02-01; First posted 2024-02-09 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Hand, Foot and Mouth Disease
MeSH Terms: conditions — Hand, Foot and Mouth Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Case cohort: Clinically diagnosed HFMD children of either sex, aged 6 months - 18 years old in the study sites
  Interventions: Diagnostic Test: PCR

INTERVENTIONS:
Diagnostic Test: PCR — PCR test for EV71, CA16, CA10, or CA6

SUMMARY:
An observational study of active case surveillance to identify the pathogens of clinically diagnosed HFMD cases aged 6 months to 18 years old recruited from puskesmas and hospitals in Indonesia.

DETAILED DESCRIPTION:
Every time suspected case of HFMD presented to the hospital, the pediatrician will inform the patient to enroll in the study. After the subject signs the informed consent, the pediatrician will give the subject designated number to enroll to the study. After gathering general information, medical history, and physical examination, the eligibility of participants will be assessed. The subject that fulfills the eligibility criteria will be enrolled in the study. All participants will collect stool sample or rectal swab to be tested with PCR test for EV71, CA (planned serotypes 16/10/6). If the result is positive, the sample will be further tested with genotype sequencing of EV71 and CoxA. For subject with respiratory symptom, skin lesion or encephalitis, extra PCR testing will be collected for PCR testing. Blood sample will also be collected from all subjects. Only 20 subjects with positive PCR result that will be tested for SVNT and PRNT. Two weeks following participant recruitment, study staff will contact the participant by phone and document the outcome of the disease as well the subject's condition.

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosed HFMD children of either sex, aged 6 months - 18 years old in the study sites
* The participant's parent/ legally accepted representative (LAR) could understand and sign a documented informed consent voluntarily before the study procedures.

Exclusion Criteria:

* NA.

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Participants with clinically diagnosed cases of HFMD will be enrolled during the epidemic season within one year or earlies.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
To identify the pathogens (EV71, CA16, CA10, and CA6) in clinically diagnosed HFMD childrenCA16, CA10, or CA6 | 12 months
  Proportions of clinically diagnosed HFMD children who are PCR- positive for EV71, CA16, CA10, or CA6

SECONDARY OUTCOMES:
To describe the clinical manifestation (symptom and severity etc.) of clinically diagnosed HFMD children | 12 months
  Distribution of HFMD symptoms and disease severity per predefined age groups, gender group (male and female), region group (urban and rural) and enterovirus type (EV71, CA16, CA10, CA6 and others) group.
To describe the genotypes of HFMD cases caused by EV71, CA16, CA10, and CA6 | 12 months
  Frequency of the genotypes of EV71, CA16, CA10 or CA6 in PCR- positive cases
To investigate role of previous infection of enterovirus EV71, coxsackie virus | 12 months
  Proportions of participants who have previous infection (SVNT, and PRNT) of EV71, Coxsackie virus

IPD SHARING:
Plan to Share IPD: Undecided